CLINICAL TRIAL: NCT04414605
Title: Oral Chinese Herbal Medicine Formula (Gu Ben Hua Yu Fang) Concurrent With Secukinumab for Severe Plaque Psoriasis
Brief Title: Oral Chinese Herbal Medicine Concurrent With Secukinumab for Severe Plaque Psoriasis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF2020-068-02
Record Dates: First submitted 2020-05-11; First posted 2020-06-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chinese herbal medicine in combination with secukinumab (Experimental): Oral Chinese herbal medicine (Gu Ben Hua Yu Fang decoction) and secukinumab will be used concurrently. The treatment duration for both secukinumab and oral Chinese herbal medicine is up to 16 weeks. Secukinumab will be administered by subcutaneous injection. The required dose (300 mg) is divided into two doses of 150 mg (contained in two separate syringes), which are injected at the same time. The first five doses (each consisting of 2 injections of 150 mg) are given at weekly intervals, with subsequent treatment given monthly (2 injections of 150 mg). Chinese herbal formula (Gu Ben Hua Yu Fang) decoction will be orally administrated twice a day. One pack of Gu Ben Hua Yu Fang will be taken for each time. Chinese herbal medicine (Gu Ben Hua Yu Fang) will not be used on the day of receiving secukinumab injection.
  Interventions: Drug: Gu Ben Hua Yu Fang decoction (Chinese herbal medicine); Drug: Secukinumab Auto-Injector [Cosentyx]

INTERVENTIONS:
Drug: Gu Ben Hua Yu Fang decoction (Chinese herbal medicine) — Chinese herbal formula (Gu Ben Hua Yu Fang) decoction will be orally administrated twice daily. One pack of Gu Ben Hua Yu Fang will be taken for each time. Chinese herbal medicine (Gu Ben Hua Yu Fang) will not be used on the day of receiving secukinumab injection.
  Other Names: Chinese herbal medicine decoction
Drug: Secukinumab Auto-Injector [Cosentyx] — Secukinumab will be administered by subcutaneous injection. The required dose (300 mg) is divided into two doses of 150 mg (contained in two separate syringes), which are injected at the same time. The first five doses (each consisting of 2 injections of 150 mg) are given at weekly intervals, with subsequent treatment given monthly (2 injections of 150 mg).
  Other Names: Cosentyx

SUMMARY:
The aim of this study is to determine whether oral Chinese herbal medicine in combination secukinumab is effective and safe in the treatment of severe psoriasis.

DETAILED DESCRIPTION:
The aim of this study is to determine whether oral Chinese herbal medicine in combination with secukinumab is effective and safe in the treatment of severe psoriasis. Eligible participants will be treated with oral Chinese herbal medicine and secukinumab concurrently. No controlled group will be set up in this trial. The primary outcome is time to relapse. Secondary outcomes include Psoriasis Area and Severity Index (PASI) 75/90, PASI score reduction rate, physician's global assessment (PGA) score, body surface area (BSA) score, visual analogue scale (VAS) score, dermatology life quality index (QLQI) and Skindex 16.

ELIGIBILITY:
Inclusion Criteria:

1. Psoriasis Area and Severity Index (PASI) score≥10
2. Meet the requirement of using secukinumab; without the history of inflammatory bowel disease (IBD)
3. Written/signed informed consent

Exclusion Criteria:

1. Unsuitable for the treatment of secukinumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Median time to relapse | Through study completion, an average of 1 year
  Median time to relapse is a time interval. The time interval will be recorded between the end of treatment and the occurrence of relapse. Relapse was defined as loss of > 50% of maximum Psoriasis Area and Severity Index (PASI) improvement compared with pretreatment baseline.

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) score | Assessment will be conducted at week 0, 1, 2, 3, 4, and every four weeks throughout the remaining period the this trial, an average of 1 year
  The improvement in Psoriasis Area and Severity Index (PASI) score from baseline after treatment; the scale scores ranged from 0-72. The higher the scores are, the more severe the patients suffer
PASI-75 | 16 weeks after treatment
  The proportion of patients who achieve at least 75% improvement in PASI score from baseline.
PASI-90 | 16 weeks after treatment
  The proportion of patients who achieve at least 90% improvement in PASI score from baseline.
Physician's global assessment (PGA) score | Assessment will be conducted on week 0, 1, 2, 3, 4, and every four weeks throughout the remaining period the this trial, an average of 1 year.
  Physician's global assessment for the condition
Pruritus Scores on the Visual Analogue Scale | Assessment will be conducted on week 0, 1, 2, 3, 4, and every four weeks throughout the remaining period the this trial, an average of 1 year.
  Pruritus will be assessed using the Visual Analogue Scales; The Scale scores ranged from 0-10; the higher the scores are, the more itching the patients suffer.
BSA | Assessment will be conducted on week 0, 1, 2, 3, 4, and every four weeks throughout the remaining period the this trial, an average of 1 year.
  the Body Surface Area
Dermatology Life Quality Index (DLQI) | Assessment will be conducted on week 0, 16 and the end of study completion (once relapse occurs, an average of 1 year).
  Questionnaire for disease-specific quality of life
Skindex16 | Assessment will be conducted on week 0, 16 and the end of study completion (once relapse occurs, an average of 1 year).
  Questionnaire for disease-specific quality of life
patients' attitudes, expectation and experience | Interview will be conducted on week 0, 16 and the end of study completion (once relapse occurs, an average of 1 year).
  Semi-structured individual interview will be conducted to explore patients' understanding and expectation for the combination therapy used in this study. Patients' experience of using the combination therapy will be recorded as well.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, PhD, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China